CLINICAL TRIAL: NCT04323878
Title: EC-COVID-PCS - Early CPAP in COVID Patients With Respiratory Failure. A Prospective Cohort Study.
Brief Title: Early CPAP in COVID-19 Patients With Respiratory Failure. A Prospective Cohort Study.
Acronym: EC-COVID-PCS
Status: Completed | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: EC-COVID-PCS-Fenice
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2021-12

CONDITIONS: Early CPAP Ventilation in COVID-19 Patients
Keywords: Early CPAP ventilation; COVID-19; Emergency Departement
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cohort study aims at prospectively collecting detailed clinical information on patients positive to or suspected of COVID-19 visiting Italian emergency departments (EDs). The objectives of the study are:

1. To monitor and describe the COVID-19 patients visiting Italian EDs.
2. To assess the prognostic impact of demographics, clinical characteristics, risk factors and pre-existing diseases.
3. To develop a predictive model, providing estimates of the prognosis using multiple relevant factors.
4. To construct a detailed database to enable comparative effectiveness research (CER), with the goal of generating hypothesis of efficacy and effectiveness of treatments, therapies and interventions, in the management and treatment of COVID-19 patients.

DETAILED DESCRIPTION:
All the ED patients positive to or suspected of COVID-19 infection will be included in the study. Descriptive reports of the collected data will be produced regularly. Different levels of aggregation will be considered: single center, province, region. In addition to providing useful elements to describe the evolution of the epidemic, the results presented in these reports will provide an accurate clinical description of a large sample of COVID-19 patients.

The study data will be leveraged to identify the most important risk factors and clinical conditions to predict poor patient outcomes. The most relevant factors will be selected using state-of-the-art techniques.

These factors will be used as predictors in multivariable predictive models, which will be developed to estimate the expected prognosis of the patients. The study outcomes will be death or need of intubation within 7 days since ED arrival and 30-day mortality. Given the dichotomous nature of these variables, the models will be developed with logistic regression. The models will be first developed when the study will enroll the minimum number of necessary patients, and periodically updated. In this way, predictive tools capable of making accurate estimates of the prognosis of patients will be returned to the clinical practice as soon as possible.

The study will record the use of treatments and drugs, such as antivirals, ACE inhibitors and sartans, whose effect on COVID-19 patients is not yet clear and mostly based on small studies. The large cohort of patients will be used to perform CER analyses and evaluate the effect of these treatments on the prognosis of patients, with appropriate statistical methodology to account for the observational nature of the data. These results will be used to refine and improve the experimental design of this project.

ELIGIBILITY:
Inclusion Criteria:

All the ED patients positive to or suspected of COVID-19 infection with at least one of the following symptoms:

* fever
* cough/dyspnea
* SpO2 < 95% in ambient air (< 91% if BPCO patient).
* positive Quick Walk Test
* respiratory symptoms or admission in ED for respiratory reason

Exclusion Criteria:

* age < 18 years
* intubated patients or patients discharged in ICU in 1 hour from ED arrival
* denied consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the ED patients positive to or suspected of COVID-19 infection with respitatory symptoms
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Death or need of intubation | 7 days since ED arrival
  The study outcomes will be death or need of intubation within 7 days since ED arrival.

SECONDARY OUTCOMES:
30-day mortality | 30 days since ED arrival
  30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Guido Bertolini, MD, Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No